CLINICAL TRIAL: NCT02239315
Title: Study of Tumor RNA Disruption Assay™ (RDA) and Its Association With a Response to Neoadjuvant Chemotherapy in Breast Cancer - A Prospective Mixed-Methods Study
Brief Title: Study of Tumor RNA Disruption Assay™ (RDA)
Acronym: RnaDx
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Murray Krahn, MD, MSc, FRCPC, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 495462
Record Dates: First submitted 2014-09-02; First posted 2014-09-12 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Breast Neoplasms
Keywords: Breast cancers; Neoadjuvant chemotherapy; RNA Disruption Assay™ (RDA) score; Pathological Complete Response (pCR); Fine Needle Aspiration Biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tumor RNA Disruption Assay™ (RDA) (Experimental): Tumor RNA Disruption Assay™ (RDA) to generate RDA score from fine needle aspiration biopsy samples of breast cancer obtained 7-14 days after the first, second and third cycles of neoadjuvant chemotherapy; and, if there is a change of chemotherapy regimen, after the first cycle of the new chemotherapy.
  Interventions: Other: Tumor RNA Disruption Assay™ (RDA)

INTERVENTIONS:
Other: Tumor RNA Disruption Assay™ (RDA) — Tumor RNA Disruption Assay™ (RDA) to generate RDA score from fine needle aspiration biopsy samples of breast cancer obtained 7-14 days after the first, second and third cycles of neoadjuvant chemotherapy; and, if there is a change of chemotherapy regimen, after the first cycle of the new chemotherapy.
  Other Names: Biomarker

SUMMARY:
The purpose of this study is to find out if the pathological complete response (pCR) to chemotherapy given before surgery (neoadjuvant chemotherapy) could be predicted by the evaluation of the RNA (ribonucleic acids) disruption pattern (RNA Disruption Assay or RDA score) obtained from a biopsy of the tumor 7 - 14 days after the first, second and third cycles of chemotherapy treatment. If we can determine the optimal time during neoadjuvant chemotherapy to measure the RDA score for the prediction of pCR, we can optimize breast cancer management.

DETAILED DESCRIPTION:
When administering neoadjuvant chemotherapy, the current practice of monitoring response to treatment is by measuring the size of the breast tumor after each cycle of chemotherapy. The drawback to this method is, it will take several weeks before we can actually measure a significant change in size; and the initial response to chemotherapy is often evident as a softening of the tumor without an apparent decrease of the tumor size. Finding a reliable way to identify early response to chemotherapy would be helpful to enable matching of chemotherapy to an individual's need.

In a previous trial of breast cancer treated with neoadjuvant chemotherapy, researchers have identified that the pCR to a full treatment of chemotherapy could be predicted by the change in RNA pattern obtained from a biopsy of the tumor half way through the chemotherapy course. [Parissenti et al. 2010] The purpose of this study is to determine if we can predict the pCR to neoadjuvant chemotherapy by examining the pattern of RNA disruption (RNA Disruption Assay or RDA score) from breast biopsy tissue obtained 7 to 14 days after the first, second and third cycle of chemotherapy. If we can determine the optimal time during neoadjuvant chemotherapy to measure the RDA score for the prediction of pCR, we can optimize breast cancer management. For example, if RDA score can identify non-responders earlier, we can switch to other chemotherapy agents and reduce the exposure to the unnecessary side-effects of ineffective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female,18 years or older;
* Able to read and write in English:
* With palpable cancer > 2cm (T2, T3) on clinical examination or clinical diagnosis of locally advanced breast cancer (LABC) (T3 or T4; or N2 or N3, according to TNM cancer staging including inflammatory breast cancer);
* Must have histological proof of breast cancer (invasive ductal or infiltrating lobular);
* Scheduled to receive neoadjuvant chemotherapy as part of their treatment plan;
* Agree to have FNAB after the first, second and third cycle of chemotherapy, and if the chemotherapy regimen is changed, an additional FNAB after the first cycle of the new chemotherapy.

Exclusion Criteria:

* Subjects who have had surgery, neoadjuvant chemotherapy or radiotherapy for the current breast cancer;
* Subjects who are pregnant or breast feeding;
* Subjects with Stage IV breast cancer;
* Psychiatric or addictive disorders that may limit the ability to give informed consent or complete the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-12; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The association between RDA score and pathological complete response (pCR) | An expected average of 6 months
  The association between tumor RDA score measured 7-14 days after the first, second and third cycles of chemotherapy and the pCR to neoadjuvant chemotherapy will be evaluated. pCR is defined as no evidence of invasive carcinoma in the breast and lymph nodes (ypT0/Tis ypN0/N0itc) on histology at the time of surgery (lumpectomy or mastectomy).

SECONDARY OUTCOMES:
The prognostic ability of RDA score | An expected average of 6 months
  The capacity of RDA score to predict pCR to neoadjuvant chemotherapy will be assessed by exploring for a cut point on the RDA score to differentiate subjects with a high likelihood of achieving pCR versus those who are less likely to achieve pCR.
The association between RDA score and clinical response (cR) | An expected average of 6 months
  The association between tumor RDA score measured 7-14 days after the first, second and third cycles of chemotherapy and clinical response to neoadjuvant chemotherapy treatment will be evaluated.
Patients' perception of fine needle aspiration biopsy (FNAB) and of breast cancer care | An expected average of 12 months
  We shall seek to understand the experiences of patients with the FNAB procedure and with the cancer care they received while participating in the study by conducting qualitative interviews of study subjects.
The cost-effectiveness of using RDA score | An expected average of 6 months
  The cost-effectiveness of using RDA score to guide neoadjuvant chemotherapy will be evaluated by measuring the cost-effectiveness of monitoring pCR to neoadjuvant chemotherapy through the RDA score and in modifying the neoadjuvant chemotherapy regimen for non-pCR patients accordingly.
The association between RDA score and Disease-Free Survival (DFS) | An expected average of 5 years
  The association between tumor RDA score measured 7-14 days after the first, second and third cycles of chemotherapy and DFS will be evaluated. DFS will be measured as the time from patient's enrollment to the event of cancer metastasis or recurrence, or death, whatever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Murray Krahn, MD,MSc,FRCPC, Principal Investigator — Director of THETA Collaborative, the F. Norman Hughes Chair in Pharmacoeconomics and Social and Administrative Pharmacy Division Head in the Faculty of Pharmacy, Professor at the University of Toronto
Locations (4):
- Canada (4):
  - Hamilton Health Sciences Juravinski Cancer Centre, Hamilton, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Sunnybrook Health Sciences Odette Cancer Centre, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Background] Parissenti AM, Chapman JA, Kahn HJ, Guo B, Han L, O'Brien P, Clemons MP, Jong R, Dent R, Fitzgerald B, Pritchard KI, Shepherd LE, Trudeau ME. Association of low tumor RNA integrity with response to chemotherapy in breast cancer patients. Breast Cancer Res Treat. 2010 Jan;119(2):347-56. doi: 10.1007/s10549-009-0531-x. PMID 19771508
- [Background] Schroeder A, Mueller O, Stocker S, Salowsky R, Leiber M, Gassmann M, Lightfoot S, Menzel W, Granzow M, Ragg T. The RIN: an RNA integrity number for assigning integrity values to RNA measurements. BMC Mol Biol. 2006 Jan 31;7:3. doi: 10.1186/1471-2199-7-3. PMID 16448564
- [Background] Guidance for Industry- Pathologic Complete Response in Neoadjuvant Treatment of High-Risk Early-Stage Breast Cancer: Use as an Endpoint to Support Accelerated Approval (May 2012). US DHHS FDA CDER; Available from: http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM305501.pdf